CLINICAL TRIAL: NCT07042113
Title: A Randomized, Open-label, Parallel-enrollment Pharmacokinetic Comparison Study of Two Formulations of Recombinant Anti-IL-4Rα Humanized Monoclonal Antibody Injection (611) Injected Subcutaneously in Healthy Adult Subjects in China
Brief Title: A Study of Two Different Formulations of 611 in Healthy Adult Subjects in China
Acronym: 611
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-611-HV-I-02
Record Dates: First submitted 2025-06-09; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tested preparation group (Experimental): Healthy subjects will receive new formulations of 611 300mg once
  Interventions: Drug: new formulations of 611
- Reference preparation group (Experimental): Healthy subjects will receive existing formulations of 611 300mg once
  Interventions: Drug: existing formulations of 611

INTERVENTIONS:
Drug: new formulations of 611 — Subjects will receive new formulations of 611 300mg once subcutaneous injection on D1
  Arms: Tested preparation group
Drug: existing formulations of 611 — Subjects will receive existing formulations of 611 300mg once subcutaneous injection on D1
  Arms: Reference preparation group

SUMMARY:
The main purpose of this study is to compare two different formulations (mixtures) of 611 in healthy participants. This study will compare how much of each formulation gets into the blood stream.

DETAILED DESCRIPTION:
This study is a randomized, open-label, parallel-designed comparative pharmacokinetic study to evaluate the biosimilarity between the formulations of 611.A total of about 180 healthy adult subjects in China were planned to be included, and the qualified subjects were randomly stratified according to the research center, body weight (≥65kg, <65kg), and randomly assigned to the test preparation group and the reference preparation group at a ratio of 1:1, and received a single subcutaneous injection of 300 mg of the experimental drug according to their group. Blood was collected on D1 and D2, D3, D4, D5, D6, D7, D8, D15, D22, D29, D43 and D57 after administration, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent for the study.
2. Male or female subjects, age 18-45 years older.
3. Within body mass index (BMI) range 19.0 to 26.0 kilograms per square meter (kg/m²).
4. The results of vital signs, physical examination, laboratory tests, electrocardiogram, chest X-ray and other examinations during the screening period are normal or judged to be abnormal by the investigator and have no clinical significance.
5. Males and females of non-childbearing potential.

Exclusion Criteria:

1. History of severe allergies or allergies to 611 and any of its components;
2. Previous or current disease that may affect the safety of the subject's participation in the trial or the in vivo process of the trial drug;
3. Any history of VKC and AKC;
4. History of drug abuse within 2 years prior to screening;
5. Alcoholism within 3 months prior to screening;
6. Those who smoke more than 5 cigarettes per day within 3 months before screening or cannot give up smoking during the period from signing the informed consent of the subject to leaving the group;
7. Those who have consumed more than 1L of strong tea, coffee and/or caffeinated beverages per day within 3 months before screening, and who have ingested chocolate or any food or drink containing caffeine, theophylline, theobromine or alcohol within 48 hours before the study administration;
8. Have active tuberculosis;
9. Presence of active infection requiring systemic treatment prior to screening or dosing;
10. Those who have used any prescription drugs, over-the-counter drugs, vitamin products or Chinese herbal medicines within 4 weeks or 5 half lives (whichever is longer) before dosing, or those who may need to receive other drugs during the trial;
11. Participated in the clinical trial of any drug or device within 3 months or 5 half-lives before dosing;
12. Receipt of any marketed or investigational biologic within 3 months or 5 half lives prior to dosing;
13. Live vaccine or live attenuated vaccine within 2 months prior to dosing or planned administration during the study;
14. Previous use of any IL-4Rα target drugs;
15. Pregnant or lactating females;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | 57 days
AUC | 57 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiangsheng
  - Shanghai General Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No